

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

# **Study Protocol**

Sponsor:

# GlaxoSmithKline Biologicals

Rue de l'Institut 89 1330 Rixensart, Belgium

# 1. PASS INFORMATION

| Title | Fluarix®/ Fluarix® Quadrivalent/ FluLaval® Quadrivalent Pregnancy Registry: a prospective, exploratory, cohort study to detect and describe abnormal pregnancy outcomes in women intentionally or unintentionally vaccinated with Fluarix® or Fluarix® Quadrivalent or FluLaval® or FluLaval® Quadrivalent during pregnancy or within 28 days preceding conception. |
|---|---|
| Protocol version identifier | 201476 (EPI-FLU-039 VS US PR) |
| Date of last version of the protocol | Final Version 1: 13 May 2014 |
| protocor | Amendment 1 Final: 27 October 2017 |
| EU PAS Register No: | Not applicable |
| Active substance | J07BB02, Influenza Virus Vaccines |
| Medicinal products: | Fluarix®, FluLaval®, Fluarix® Quadrivalent, FluLaval® Quadrivalent, Inactivated Influenza Virus Vaccines |
| Product reference: | Not applicable |
| Procedure number: | Not applicable |
| Marketing Authorization<br>Holder | GlaxoSmithKline Biologicals Rue de l'Institut 89 |
| | 1330 Rixensart, Belgium |
| Joint PASS | No |
| Research question and objectives | To describe the characteristics of prospectively reported pregnancies (women vaccinated with <i>Fluarix</i> or <i>FluLaval</i> or <i>Fluarix Quadrivalent</i> or <i>FluLaval Quadrivalent</i> during pregnancy or |

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

| | Protocol Amendment 1 Final |
|---|---|
| | within 28 days preceding conception) with abnormal pregnancy outcomes. |
| | To assess the proportion of prospectively reported pregnancies (women vaccinated with <i>Fluarix</i> or <i>FluLaval</i> or <i>Fluarix Quadrivalent</i> or <i>FluLaval Quadrivalent</i> during pregnancy or within 28 days preceding conception) with abnormal pregnancy outcomes. |
| <b>Country of study</b> | United States |
| Authors (Amended on 27<br>October 2017) | Coordinating author: |
| · | • XPE Pharma & Science, contractor for GSK Biologicals |
| | GSK contributors: |
| | Director, Safety Evaluation & Risk Management, Vaccine Clinical Safety and Pharmacovigilance |
| | <ul> <li>PPD , Director, Safety Evaluation</li> <li>&amp; Risk Management, Vaccine Clinical</li> <li>Safety and Pharmacovigilance</li> </ul> |
| | Director and Head, Clinical Safety Sciences, Vaccine Clinical Safety and Pharmacovigilance |
| | VP, Head Vaccine Clinical Safety and Pharmacovigilance |
| | Director, Global Clinical R&D |
| | Senior Manager, Vaccine Value & Health Science Epidemiology |
| | PPD , Director, Vaccine Value & Health Science Epidemiology |
| | Senior Manager, Regulatory Affairs |
| | • PPD , Safety Scientist, |
| | Safety Evaluation & Risk Management, Vaccine Clinical Safety and Pharmacovigilance |
| | • PPD , Head, Safety Evaluation & Risk Management, Vaccine Clinical Safety and Pharmacovigilance |

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final



# 2. MARKETING AUTHORIZATION HOLDER

| Marketing authorization holder | GlaxoSmithKline Biologicals |
|---|---|
| | Rue de l'Institut 89, 1330 Rixensart, Belgium |
| | , , , |

© [2014-2017] GSK group of companies or its licensor

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | PASS | INFORM | ATION | 1 |
| 2. | MARK | ETING A | UTHORIZATION HOLDER | 3 |
| LIS | T OF A | BBREVIA | TIONS | 8 |
| 3. | RESP | ONSIBLE | PARTIES | 9 |
| 4. | ABST | RACT | | 9 |
| 5. | AMEN | IDMENTS | S AND UPDATES | 13 |
| 6. | MILES | STONES ( | (AMENDED ON 27 OCTOBER 2017) | 13 |
| 7. | RATIC<br>7.1. | Backgro<br>7.1.1. | ND BACKGROUNDund Trivalent influenza vaccines | 14<br>15<br>16 |
| | | 7.1.2.<br>7.1.3.<br>7.1.4. | Quadrivalent influenza vaccines 7.1.2.1. Animal studies 7.1.2.2. Post marketing exposure in pregnant women 7.1.2.3. GSK sIIVs Medical conditions for use (Amended on 27 October 2017). Characteristics of exposure. | 17<br>18<br>19 |
| | 7.2. | 7.1.5.<br>Rational | Potential benefits of producte | |
| 8. | RESE<br>8.1. | | JESTION AND OBJECTIVESary objectives | |
| 9. | RESE<br>9.1. | | ETHODS esign Overview (Amended on 27 October 2017) Rationale for study design | 20<br>20 |
| | 9.2. | Setting .<br>9.2.1. | Study population | 22<br>22 |
| | | 9.2.2.<br>9.2.3.<br>9.2.4.<br>9.2.5.<br>9.2.6. | 9.2.1.2. Potential annual exposure (Amended on 27 October 2017) | 22<br>22<br>23<br>23 |
| | 9.3. | | SPrimary endpoint | 23<br>23 |

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

| | | | | 1 Totocol 7 till oli dillion | |
|---|---|---|---|---|---|
| | | | 9.3.2.1. | Questionnaire for initial data collection | |
| | | | | (Amended on 27 October 2017) | 24 |
| | | | 9.3.2.2. | Questionnaire for pregnancy outcome data | |
| | | | | collection (Amended on 27 October 2017) | |
| | | | 9.3.2.3. | Questionnaire for infant data collection | |
| | 9.4. | | | nded on 27 October 2017) | |
| | 9.5. | | | | |
| | 9.6. | | 0 | | |
| | | 9.6.1. | | ction (Amended on 27 October 2017) | |
| | | 9.6.2. | | g of reports (Amended on 27 October 2017) | 26 |
| | | | 9.6.2.1. | Solicitation of outcomes (Amended on 27 | |
| | | | | October 2017) | 27 |
| | | | 9.6.2.2. | Classification of outcomes | |
| | 9.7. | | | ended on 27 October 2017) | |
| | 9.8. | Quality of | control | | 29 |
| | 9.9. | Limitatio | ns of the re | search methods | 30 |
| 10. | | | | I SUBJECTS | 30 |
| | 10.1. | | | cal considerations, including the informed | |
| | | consent | process | | 30 |
| | | 0 E M E M E | | ODTING OF ADVEDOR EVENTO (ADVEDOR | |
| 11. | | | | ORTING OF ADVERSE EVENTS/ADVERSE | 0.4 |
| | REAC | HONS | | | 31 |
| 40 | DI ANG | COD DI | CCENTINIAT | THE AND COMMUNICATING STUDY | |
| 12. | | | | ING AND COMMUNICATING STUDY | 24 |
| | KE201 | _15 (AMI | ENDED OF | N 27 OCTOBER 2017) | 31 |
| 12 | DEEE | DENICES | | | 21 |
| ı٥. | | ILINGES. | | | ۱ |

# 201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

# **LIST OF TABLES**

| | P | AGE |
|---|---|---|
| Table 1 | Current Pregnancy Registry Protocols being conducted for Fluarix, FluLaval, Fluarix Quadrivalent and FluLaval Quadrivalent | 14 |
| Table 2 | Outcomes of pregnancy exposed to Fluarix | 16 |
| Table 3 | Outcomes of pregnancy exposed to FluLaval | 17 |
| Table 4 | Outcomes of pregnancy exposed to Fluarix Quadrivalent | 18 |
| Table 5 | Year of initial US approval for GSK sIIVs | 19 |

# 201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

# **LIST OF ANNEXES**

| | | PAGE |
|---------|-------------------------------------------------------|------|
| ANNEX 1 | List of stand-alone documents | 34 |
| ANNEX 2 | ENCePP Checklist for study protocols | 35 |
| ANNEX 3 | Glossary of terms | 36 |
| ANNEX 4 | Amendments and administrative changes to the protocol | 38 |
| ANNEX 5 | Trademarks | 57 |
| ANNEX 6 | Protocol Amendment 1 sponsor signatory approval | 58 |

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

## LIST OF ABBREVIATIONS

**ACIP** Advisory Committee on Immunization Practices

**AE** Adverse Event

**BLA** Biologics License Application

**CBER** Center for Biologics Evaluation and Research

CDC Centers for Disease Control and Prevention

**EDD** Estimated Date of Delivery

**FDA** Food and Drug Administration

**GCP** Good Clinical Practice

**GSK** GlaxoSmithKline

**HA** Hemagglutinin

**HCP** Healthcare Professional

**ICH** International Conference on Harmonization

IM Intramuscular

IND Investigational New Drug

LMP Last Menstrual Period

MACDP Metropolitan Atlanta Congenital Defects Program

**PASS** Post Authorization Safety Study

PI Prescribing Information

sIIV(s) seasonal Inactivated Influenza Vaccine(s)

US United States

VCSP Vaccine Clinical Safety and Pharmacovigilance

## 3. RESPONSIBLE PARTIES

GlaxoSmithKline (GSK) Biologicals has the overall responsibility for the conduct of the study.

## 4. ABSTRACT

**Title** 

Fluarix®/ FluLaval®/ Fluarix® Quadrivalent/ FluLaval® Quadrivalent Pregnancy Registry: an exploratory prospective, cohort study to detect and describe abnormal pregnancy outcomes in women intentionally or unintentionally vaccinated with Fluarix® or Fluarix® Quadrivalent or FluLaval® or FluLaval® Quadrivalent during pregnancy or within 28 days preceding conception.

201476 (EPI-FLU-039 VS US PR), Amendment 1 Final: 27 October 2017

Main author

PPD , Director, Safety Evaluation & Risk Management, Vaccine Clinical Safety and Pharmacovigilance, GSK Biologicals

Rationale and background

The four seasonal Inactivated Influenza Vaccines *Fluarix*, *FluLaval*, *Fluarix Quadrivalent* and *FluLaval Quadrivalent* (collectively referred to as GSK seasonal Inactivated Influenza Vaccines [GSK sIIVs]) are approved in the United States (US) for prevention of disease caused by influenza A subtype viruses and type B viruses contained in the vaccine in persons 3 years of age and older. Pregnant women may inadvertently be vaccinated with GSK sIIVs during the first trimester, before pregnancy is known. In general, the women are closely monitored throughout the remainder of the pregnancy.

The purpose of this pregnancy registry study is to detect and describe abnormal pregnancy outcomes in women intentionally or unintentionally vaccinated with GSK sIIVs. The combination of the large number of women who are of reproductive capacity in the indicated age range for vaccination with these vaccines and the lack of data concerning vaccination with GSK sIIVs during pregnancy makes such a Registry an important component of the ongoing program to assess the safety of these four vaccines. The intent of the Registry is to prospectively collect data such as vaccination with GSK sIIVs during pregnancy or within 28 days preceding conception, potential confounding factors (such

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

as exposure to other medications) and information related to the outcome of the pregnancy.

# Research question and objectives

## **Co-primary objectives**

- To describe the characteristics of prospectively reported pregnancies (women vaccinated with *Fluarix* or *FluLaval* or *Fluarix Quadrivalent* or *FluLaval Quadrivalent* during pregnancy or within 28 days preceding conception) with abnormal pregnancy outcomes.
- To assess the proportion of prospectively reported pregnancies (women vaccinated with *Fluarix* or *FluLaval* or *Fluarix Quadrivalent* or *FluLaval Quadrivalent* during pregnancy or within 28 days preceding conception) with abnormal pregnancy outcomes.

## Study design (Amended on 27 October 2017)

- This study is a transition of existing ongoing pregnancy registries for Fluarix, FluLaval and Fluarix Quadrivalent and an ongoing PASS for FluLaval Quadrivalent into a combined PASS for these four GSK sIIVs
- This is an exploratory prospective, observational, cohort study. The GSK sIIVs pregnancy registry study requires voluntary, prospective\* reporting of eligible pregnancies by patients and healthcare professionals (HCPs). Data such as vaccination with GSK sIIVs during pregnancy or within 28 days preceding conception, potential confounding factors (such as exposure to other medications) and information related to the outcome of the pregnancy will be collected prospectively.

\*Some pregnancy exposures may be reported when the outcome is unknown (prospective reports).

Some pregnancy exposures may be reported after pregnancy outcome has been identified (retrospective reports). The Registry will capture retrospective reports, but these reports will not be included in the analyses of prospective reports.

- This study is a post-marketing commitment in the US.
- Study population: pregnant women, vaccinated with GSK sIIVs during pregnancy or within 28 days preceding conception volunteering to take part in the study.
- Type of study: self-contained.
- Data collection: Initial and follow-up data will be collected using questionnaires (*Initial notification* form, *Pregnancy outcome* form *and 6 and 12-month post-*

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

delivery follow-up form). Initial data can be collected from pregnant subjects, their healthcare providers or both. Follow-up of cases is performed within 2 months of the estimated date of delivery (EDD) to ascertain outcome and approximately 6 months and 12 months after the EDD (for all live births for whom the contact details of their HCP will be available) to ascertain the presence of birth defects not diagnosed before. Follow-up questionnaires can only be completed by healthcare providers and/or HCP staff.

 After transition of the ongoing pregnancy registries into one combined PASS for GSK sIIVs, data will be collected for a minimum of 5 years starting Q2 2014

Population, including the setting and study population (Amended on 27 October 2017) In the US, GSK sIIVs are indicated for prevention of disease caused by influenza A subtype viruses and type B viruses contained in the vaccine. Currently, GSK sIIVs are approved for use in persons 3 years of age and older or 6 months of age and older, depending on the vaccine.

#### Size of the potential "at-risk" population

In the year 2012, the fertility rate in the US was 63.2 births per 1000 women aged 15-44 years and there were 3.96 million births [CDC, 2012].

#### Number of pregnant vaccinees

Although the number of pregnant women who will be vaccinated with GSK IIVs *through this registry* is impossible to predict, experiences with other vaccine pregnancy registries indicate that it is likely that fewer than 100 pregnancies per year will be registered for each of the vaccines.

#### Variables

#### **Primary endpoint**

Occurrence of abnormal pregnancy outcomes in women intentionally or unintentionally vaccinated with GSK sIIVs during pregnancy or within 28 days preceding conception.

Data sources (Amended on 27 October 2017) Reporting of vaccine-exposed pregnancies to the Registry is voluntary. Registration can be initiated from a HCP or from a consumer. Permission *from consumers* is requested to obtain confirmation and follow-up from their HCP, *as well as follow-up from the HCP of their infant*. A toll-free telephone number for reporting adverse events (AEs) and vaccine-exposed pregnancies to the Registry are listed in the product information leaflet and on the GSK Registry website.

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

Retrospective post-marketing reports and relevant scientific publications are potential sources of additional information.

Study size

No minimum sample size is required for this descriptive, exploratory study.

Please refer to Abstract Section "Study population" above for the size of the potential "at-risk" population and the number of pregnant vaccinees.

Data analysis (Amended on 27 October 2017) Pregnancy outcomes include spontaneous abortion (pregnancy loss before 22 weeks gestation), fetal deaths/stillbirths (loss at or after 22 weeks gestation), elective/therapeutic abortions and live births. The presence or absence of birth defects or other abnormalities is evaluated within each of the preceding outcome categories.

Pregnancy outcomes are stratified by the trimester of exposure, with an additional stratum for preconception exposure with no subsequent administration of vaccine during pregnancy. Reports of multiple exposures during a pregnancy are classified by the earliest trimester of exposure. The calculations of risk for birth defects are made by dividing the number of infants with birth defects by the total number of infants with and without birth defects. An exact 95% confidence interval is calculated using standard statistical software. The outcomes of the study will be assessed against known rates from an external reference group for the likelihood of a safety signal warranting further investigation.

Spontaneous abortions without birth defects are excluded from the risk calculations.

All defects regardless of trimester of vaccine exposure will be included in the periodic summary reports of this Registry and stratified by trimester of exposure.

A section of each periodic summary report, separate from the analysis of prospective reports, will describe all abnormal outcomes of retrospectively reported cases.

Milestones (Amended on 27 October 2017) Summary reports with cumulative analyses will be written annually and submitted with the Periodic Benefit-Risk Evaluation Report (PBRER) for each GSK sIIV. A final report will be written and submitted approximately 18 months after the last annual report.

After submission of the final report, GSK will continue the Registry pending Center for Biologics Evaluation and

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

Research (CBER) review of the report and determination

whether the Registry can be discontinued.

**References** Centers for Disease Control and Prevention (CDC). Recent

Trends in Births and Fertility Rates Through December 2012.

Available at

http://www.cdc.gov/nchs/data/hestat/births fertility december 2

012/births fertility december 2012.htm

Accessed 29 August 2013.

## 5. AMENDMENTS AND UPDATES

The summary of the amendment is provided in ANNEX 4

# 6. MILESTONES (AMENDED ON 27 OCTOBER 2017)

| Milestone | Planned date <sup>a</sup> |
|----------------------------------------------|---------------------------|
| Start of data collection | 01 June 2014 <sup>b</sup> |
| End of data collection | 31 May 2019 ° |
| Annual report 1 (2014-2015 influenza season) | 10 February 2016 |
| Annual report 2 (2015-2016 influenza season) | 10 February 2017 |
| Annual report 3 (2016-2017 influenza season) | 10 February 2018 |
| Annual report 4 (2017-2018 influenza season) | 10 February 2019 |
| Annual report 5 (2018-2019 influenza season) | 10 February 2020 |
| Final report | August 2021 |

<sup>&</sup>lt;sup>a</sup> The *Fluarix* and *FluLaval* Registries were originally initiated on 02 Sep 2011. The *Fluarix Quadrivalent* and *FluLaval Quadrivalent* Registries were originally initiated on 30 Aug 2013 and 30 Nov 2013, respectively. *In* **2014**. the ongoing Registries **were** combined and converted into a PASS. GSK plans to continue the Registry for a minimum of 5 years, starting Q2 2014.

<sup>&</sup>lt;sup>b</sup> Women vaccinated with GSK sIIVs during pregnancy or within 28 days preceding conception, reported before the planned date of start of data collection (01 June 2014) but for which the pregnancy outcome is not yet known, may be enrolled retroactively in the Registry.

c After submission of the final report, GSK will continue the Registry pending Center for Biologics Evaluation and Research (CBER) review of the report and determination whether the Registry can be discontinued.

#### 7. RATIONALE AND BACKGROUND

## 7.1. Background

Both *Fluarix* and *Fluarix Quadrivalent* vaccines are manufactured by GSK Biologicals, in Dresden, Germany.

Both *FluLaval* and *FluLaval Quadrivalent* vaccines are manufactured by ID Biomedical Corporation of Quebec, a subsidiary of GSK; in Quebec City, Canada.

GSK currently has 4 Pregnancy Registry protocols that have been submitted to Investigational New Drug (IND) and Biologics License Applications (BLAs). These were submitted either as a postmarking commitment or as voluntary pharmacovigilance activities in a Risk Management Plan for the GSK sIIVs. See Table 1 for information on these registries.

Table 1 Current Pregnancy Registry Protocols being conducted for *Fluarix*, *FluLaval*, *Fluarix Quadrivalent* and *FluLaval Quadrivalent* 

| Product Name | File Number | Submission Date of<br>Pregnancy Registry<br>Protocol | Registry Starting<br>Date |
|---|---|---|---|
| Fluarix | 125127 | 31 August 2010 (Sequence<br>No. 0065) | 02 September<br>2011 |
| FluLaval | 125163/181 | 10 August 2010 (Sequence<br>No. 0027) | 02 September<br>2011 |
| Fluarix<br>Quadrivalent | 125127<br>BB-IND 114473 | 15 April 2013 (Sequence<br>No. 0181)<br>13 June 2013 (Sequence<br>No. 0036) | 30 August 2013 |
| FluLaval<br>Quadrivalent | 125163<br>BB-IND 14466 | 29 October 2013 (Sequence<br>No. 0157)<br>28 October 2013 (Sequence<br>No.0032) | 30 November 2013 |

## 7.1.1. Trivalent influenza vaccines

Fluarix and FluLaval are both split virion, inactivated influenza vaccines consisting of equal amounts of three monovalent viral antigen bulks prepared from influenza strains A/H1N1, A/H3N2 and one B strain. One dose of the split inactivated vaccine contains 15 μg hemagglutinin (HA) for each of the three influenza virus strains, for a total of 45 μg HA/0.5 mL dose.

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

#### 7.1.1.1. Animal studies

Animal reproduction studies were performed in female rats using 0.1 mL (approximately 56 times the human dose based on average weight) of *Fluarix* administered 28 days before mating and on Days 6, 8, 11 and 15 of gestation. There were no adverse effects on mating performance or fertility of the female rats, and no adverse effects on embryo/fetal survival, growth or development, or the pre- or post-natal survival, growth or development of the offspring up to 25 days of age [Fluarix Prescribing Information (PI), 2013].

In a reproductive and developmental toxicity study, the effects of *FluLaval* on embryofetal and pre-weaning development were evaluated in pregnant rats. Animals were administered *FluLaval* by intramuscular injection, once prior to gestation and on gestation days 6, 8, 11, and 15 during the period of organogenesis, at a dose of 0.1 mL/rat/occasion (approximately 40-fold excess relative to the projected human dose on a body weight basis). No adverse effects on mating, female fertility, pregnancy, parturition, lactation parameters, and embryo-fetal or pre-weaning development were observed. There were no vaccine-related fetal malformations or other evidence of teratogenesis [FluLaval PI, 2013].

## 7.1.1.2. Post marketing exposure in pregnant women

#### Fluarix:

Overall, as of 31 *May 2017*, GSK had received *236* reports of exposure to *Fluarix* during pregnancy since its launch on 04 July 1991. The outcomes of the *236* pregnancies are summarized in Table 2.

Table 2 Outcomes of pregnancy exposed to *Fluarix* 

| Outcome | Number of Cases since launch (n) |
|---|---|
| Live infant, no apparent congenital anomaly * | 52 |
| Live infant with congenital anomaly | 1 |
| Elective termination, no apparent congenital anomaly * | 0 |
| Elective termination with congenital anomaly | 1 |
| Spontaneous abortion, no apparent congenital anomaly * | 8 |
| Spontaneous abortion with congenital anomaly | 1 |
| Stillbirth, no apparent congenital anomaly * | 0 |
| Stillbirth with congenital anomaly | 0 |
| Ectopic pregnancy | 0 |
| Molar pregnancy | 0 |
| Pregnancy ongoing, lost to follow-up or unknown | 173 |
| Total | 236 |

<sup>\*</sup> Pregnancy outcome categories stating no apparent congenital anomaly include outcomes where it is unknown whether a congenital anomaly occurred.

#### FluLaval:

Overall, as of 31 May 2017, GSK had received 130 reports of exposure to FluLaval during pregnancy since launch on 18 December 1992. The outcomes of the 130 pregnancies are summarized in Table 3.

Table 3 Outcomes of pregnancy exposed to FluLaval

| Outcome | Number of Cases since launch |
|---|---|
| Live Infant, no apparent congenital anomaly * | 46 |
| Live infant with congenital anomaly | 1 |
| Elective termination, no apparent congenital anomaly* | 0 |
| Elective termination with congenital anomaly | 0 |
| Spontaneous abortion, no apparent congenital anomaly* | 3 |
| Spontaneous abortion with congenital anomaly | 0 |
| Stillbirth, no apparent congenital anomaly* | 0 |
| Stillbirth with congenital anomaly | 0 |
| Ectopic pregnancy | 0 |
| Molar pregnancy | 0 |
| Pregnancy ongoing / Unknown / Lost to Follow-up | 80 |
| Total | 130 |

<sup>\*</sup> Pregnancy outcome categories stating no apparent congenital anomaly include outcomes where it is unknown whether a congenital anomaly occurred.

#### 7.1.2. Quadrivalent influenza vaccines

Fluarix Quadrivalent and FluLaval Quadrivalent are split virion, inactivated influenza vaccines consisting of equal amounts of four monovalent viral antigen bulks prepared from influenza strains A/H1N1, A/H3N2 and two B strains (one B/Yamagata lineage and one B/Victoria lineage). One dose of the split inactivated vaccine contains 15 μg HA for each of the four influenza virus strains, for a total of 60 μg HA/0.5 mL dose.

#### 7.1.2.1. Animal studies

Reproductive and developmental toxicity of *Fluarix Quadrivalent* and *FluLaval Quadrivalent* has been studied in female rats at doses approximately 80 times the human dose (on a mg/kg basis) and no evidence of impaired female fertility or harm to the fetus was observed.

In reproductive and developmental toxicity studies, the effect of *Fluarix Quadrivalent* and *FluLaval Quadrivalent* on embryo-fetal and pre-weaning development was evaluated in rats. Animals were administered *Fluarix Quadrivalent* or *FluLaval Quadrivalent* by intramuscular (IM) injection twice prior to gestation, during the period of organogenesis (gestation days 3, 8, 11 and 15) and during lactation (day 7), 0.2 mL/rat/occasion (approximately 80-fold excess relative to the projected human dose on a body weight basis). No adverse effects on embryo-fetal or peri- and post-natal development, no

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

maternal toxicity and no impact on F<sub>0</sub> female clinical condition, food consumption, body weight, mating performance, fertility or ability to produce a live litter were observed during these studies [Fluarix Quadrivalent PI, 2013; FluLaval Quadrivalent PI, 2013].

#### 7.1.2.2. Post marketing exposure in pregnant women

Fluarix Quadrivalent:

Overall, as of 31 May 2017, GSK had received 64 reports of exposure to Fluarix Quadrivalent during pregnancy since launch on 5 August 2013. The outcomes of the 64 pregnancies are summarized in Table 4.

Table 4 Outcomes of pregnancy exposed to Fluarix Quadrivalent

| Outcome | Number of Cases<br>since launch (n) |
|---|---|
| Live infant, no apparent congenital anomaly * | 15 |
| Live infant with congenital anomaly | 0 |
| Elective termination, no apparent congenital anomaly * | 0 |
| Elective termination with congenital anomaly | 0 |
| Spontaneous abortion, no apparent congenital anomaly * | 1 |
| Spontaneous abortion with congenital anomaly | 1 |
| Stillbirth, no apparent congenital anomaly * | 0 |
| Stillbirth with congenital anomaly | 0 |
| Ectopic pregnancy | 0 |
| Molar pregnancy | 0 |
| Pregnancy ongoing, lost to follow-up or unknown | 47 |
| Total | 64 |

FluLaval Quadrivalent:

Overall, as of 31 May 2017, GSK had received 8 reports of exposure to FluLaval Quadrivalent during pregnancy since launch on 15 August 2013. At the time of the reporting, all 8 pregnancies were ongoing or lost to follow-up.

#### 7.1.2.3. GSK sIIVs

Animal studies did not reveal any developmental or reproductive safety issue for GSK sIIVs. There are, however, no adequate and well-controlled studies of these vaccines in pregnant women. Review of the collective post marketing exposure experience of GSK sIIVs does not suggest a safety signal. It is not known whether GSK sIIVs can have negative effects on human reproductive capacity or pregnancy

outcomes. It is generally accepted that inactivated vaccines pose no risk to the pregnant or lactating women (Centers for Disease Control and Prevention [CDC, 2002]).

## 7.1.3. Medical conditions for use (Amended on 27 October 2017)

The GSK sIIVs are approved by the US Food and Drug Administration (FDA) for prevention of disease caused by influenza A subtype viruses and type B viruses contained in the vaccines (Table 5). In the US, the GSK sIIVs are approved for use in persons 3 years of age and older or 6 months of age and older, depending on the vaccine.

Table 5 Year of initial US approval for GSK sllVs

| GSK sllV | Initial US Approval |
|-----------------------|---------------------|
| Fluarix | 2005 |
| FluLaval | 2006 |
| Fluarix Quadrivalent | 2012 |
| FluLaval Quadrivalent | 2013 |

## 7.1.4. Characteristics of exposure

Pregnant women may inadvertently be vaccinated with GSK sIIVs during the first trimester, before pregnancy is known. In general, the women are closely monitored throughout the remainder of the pregnancy.

Refer to Section 9.2.1.2 for potential annual exposure in pregnant women.

## 7.1.5. Potential benefits of product

Because of the increased rate of hospitalization for serious complications of influenza among pregnant women, particularly in the third trimester [Neuzil, 1998], the CDC Advisory Committee on Immunization Practices (ACIP) recommends that any woman who will be pregnant during the influenza season should be vaccinated for influenza [CDC, 2011] and the American College of Obstetrics and Gynecology guidelines indicate that pregnant women may be vaccinated with IIV during any trimester [ACOG, 2004].

#### 7.2. Rationale

The purpose of this pregnancy registry study is to detect and describe abnormal pregnancy outcomes in women intentionally or unintentionally vaccinated with any of the four GSK sIIVs. The combination of the large number of women who are of reproductive capacity in the indicated age range for vaccination with GSK sIIVs, and the lack of data concerning vaccination during pregnancy, makes such a Registry an important

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

component of the ongoing program to assess the safety of these vaccines. This study is a transition of existing ongoing pregnancy registries for *Fluarix*, *FluLaval*, and *Fluarix Quadrivalent* and an ongoing PASS for *FluLaval Quadrivalent* into a combined PASS for GSK sIIVs.

The Registry requires voluntary, prospective reporting of eligible pregnancies by patients and healthcare professionals (HCPs). Patient confidentiality is strictly maintained. The intent of the Registry is to prospectively collect data such as vaccination with any of the four GSK sIIVs during pregnancy or within 28 days preceding conception, potential confounding factors (such as exposure to other medications) and information related to the outcome of the pregnancy.

The GSK sIIV pregnancy registry study will be maintained by GSK's Vaccine Clinical Safety and Pharmacovigilance (VCSP) department.

## 8. RESEARCH QUESTION AND OBJECTIVES

## 8.1. Co-primary objectives

- To describe the characteristics of prospectively reported pregnancies (women vaccinated with *Fluarix* or *FluLaval* or *Fluarix Quadrivalent* or *FluLaval Quadrivalent* during pregnancy or within 28 days preceding conception) with abnormal pregnancy outcomes.
- To assess the proportion of prospectively reported pregnancies (women vaccinated with *Fluarix* or *FluLaval* or *Fluarix Quadrivalent* or *FluLaval Quadrivalent* during pregnancy or within 28 days preceding conception) with abnormal pregnancy outcomes.

Refer to Section 9.3.1 for the definition of the primary endpoint.

#### 9. RESEARCH METHODS

## 9.1. Study design

## 9.1.1. Overview (Amended on 27 October 2017)

- This study is a transition of existing ongoing pregnancy registries for *Fluarix*, *FluLaval*, and *Fluarix Quadrivalent* and an ongoing PASS for *FluLaval Quadrivalent* into a combined PASS for GSK sIIVs.
- This is an exploratory, prospective, observational, cohort study.
- The GSK sIIV pregnancy registry study requires voluntary, prospective\* reporting of eligible pregnancies by patients and HCPs. Data such as vaccination with a GSK sIIV during pregnancy or within 28 days preceding conception, potential confounding factors (such as exposure to other medications) and information related to the outcome of the pregnancy will be collected prospectively.

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

\*Some pregnancy exposures may be reported when the outcome is unknown (prospective reports).

Some pregnancy exposures may be reported after pregnancy outcome has been identified (retrospective reports). The Registry will capture retrospective reports, but these reports will not be included in the analyses of prospective reports.

- This study is a post-marketing commitment in the US.
- Study population: pregnant women, vaccinated with GSK sIIV during pregnancy or within 28 days preceding conception, volunteering to take part in the study.
- Type of study: self-contained.
- Data collection: initial and follow-up data will be collected using 3 questionnaires. Data for enrollment will be collected using the Initial Notification Form. Follow-up of cases is performed within 2 months of the estimated date of delivery (EDD) to ascertain pregnancy outcome (through the Pregnancy Outcome Form) and approximately 6 months and 12 months after the EDD (for all live births for whom the contact details of their HCP will be available) to ascertain the presence of birth defects not diagnosed before (through the 6- and 12-month post-delivery Follow-Up Form).
- After transition of the ongoing pregnancy registrations into one combined PASS for GSK sIIVs, data will be collected for a minimum of 5 years starting Q2 2014.

## 9.1.2. Rationale for study design

This is a *condition based* Registry *as opposed to a disease registry*. After market authorization, adverse events (AEs) that occur after administration of the vaccine can and should always be reported. In that case, however, there is no clear group in which the events occur and so a proper rate of occurrence cannot be estimated. In this pregnancy registry, participants are recruited between administration of the vaccine and the potential occurrence of an AE (i.e., a teratogenic effect in the offspring). This allows for a more proper estimation of the rate of occurrence of these events. Nevertheless, the results of this study still need to be regarded with caution as the exact number of women exposed during pregnancy is unknown. Incidences of events cannot therefore be calculated from the study data.

Furthermore, it is likely that pregnant women who accept vaccination may differ from those who refuse vaccination in underlying health status, propensity to seek medical care, propensity to report AEs and differences in access to medical care in general. The differential response/participation by vaccinated versus unvaccinated pregnant women in a pregnancy registry could significantly bias risk estimates and possibly in unpredictable ways, because of the inability to collect adequate data to characterize the non-responders. Therefore, the risks of any identified birth defects will be compared to those in the general population, such as that defined by the Metropolitan Atlanta Congenital Defects Program (MACDP).

## 9.2. Setting

## 9.2.1. Study population

#### 9.2.1.1. Patient population (Amended on 27 October 2017)

In the US, the GSK sIIVs are indicated for prevention of disease caused by influenza A subtype viruses and type B viruses contained in the vaccine. GSK sIIVs are approved for use in persons 3 years of age and older or 6 months of age and older, depending on the vaccine.

The study population includes women vaccinated with any of the four GSK sIIVs during pregnancy or within 28 days preceding conception.

## 9.2.1.2. Potential annual exposure (Amended on 27 October 2017)

#### Size of the potential "at-risk" population

In the year 2012, the fertility rate in the US was 63.2 births per 1000 women aged 15-44 years and there were 3.96 million births [CDC, 2012].

## Number of pregnant vaccinees

The four GSK sIIVs are classified as Pregnancy Category B. Although the number of pregnant women who will be vaccinated with GSK sIIV *with this registry* is impossible to predict, experiences with other vaccine pregnancy registries (e.g., smallpox vaccine [CDC, 2003], varicella vaccine [Shields, 2001] and *Twinrix*) indicate that it is likely that fewer than 100 pregnancies per year will be registered for each of the vaccines.

#### 9.2.2. Patient recruitment (Amended on 27 October 2017)

Reporting of vaccine-exposed pregnancies to the Registry is voluntary. Reporters become aware of the Registry through the US Prescribing Information (PI) and, *in the case of healthcare providers*, the GSK Registry website. The PIs for each of the sIIVs and GSK *Registry* website each give a brief summary of the purpose and intent of the Registry, along with contact information. *The forms for enrolling and reporting outcomes are also accessible to healthcare providers through the GSK Registry website*.

Additionally, GSK has requested that information regarding GSK pregnancy registries be posted directly on the FDA website.

#### 9.2.3. Selection of a comparison group

This registry study is a prospective cohort study. Active enrollment of a valid internal comparison group is not possible. The outcomes of the study will be assessed against known rates from an external reference group for the likelihood of a safety signal warranting further investigation. Background risks from existing, external systems (e.g., the National Birth Defects Prevention Network and the National Center for Health Statistics) will be used.

## 9.2.4. Study period

GSK proposes to continue the Registry for a minimum of 5 years (5 influenza seasons), starting in Q2 2014. Enrollment is planned to take place during the following Northern Hemisphere influenza seasons: 2014-15, 2015-16, 2016-17, 2017-18 and 2018-19. After submission of the final report, GSK will continue the Registry pending CBER review of the report and determination whether the Registry can be discontinued.

#### 9.2.5. Inclusion criteria (Amended on 27 October 2017)

A subject will be included in the Registry if all of the following criteria are met:

- Exposure to GSK sIIVs occurs during pregnancy or within 28 days preceding conception.
- Subject is a US resident.
- A HCP is identified (name, address and phone number).
- Subject can be identified (by GSK or HCP).

Data from registered subjects will be included in the analyses if the following criterion is met:

• Pregnancy is ongoing and the outcome is unknown at the time of initial report.

#### 9.2.6. Exclusion criterion

Data from registered subjects will not be included in the analyses if the following criterion is met:

• Outcome of pregnancy is known at the time of initial report. Types of known outcomes include prenatal testing reports in which the results are abnormal or outside the reference range, indicating possible abnormality in the fetus.

#### 9.3. Variables

## 9.3.1. Primary endpoint

• Occurrence of abnormal pregnancy outcomes in women intentionally or unintentionally vaccinated with *Fluarix* or *FluLaval* or *Fluarix Quadrivalent* or *FluLaval Quadrivalent* during pregnancy or within 28 days preceding conception.

## 9.3.2. Data to be collected (Amended on 27 October 2017)

Data will be collected using 3 questionnaires; one for enrollment (i.e. Initial Notification Form), one for follow-up data after the EDD (i.e. Pregnancy Outcome Form) and one for infant data at about 6 and 12 months after EDD (i.e. 6- and 12-month post-delivery Follow-Up Form).

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

# 9.3.2.1. Questionnaire for initial data collection (Amended on 27 October 2017)

The following data will be collected using the questionnaire for initial data collection (i.e. *Initial Notification Form*):

- Patient identifier.
- Maternal medical and family history including date of birth, date of last menstrual period (LMP), EDD, ethnicity.
- Type of conception.
- Prenatal testing.
- Number and outcome of previous pregnancies, including details of birth defects if applicable.
- Maternal/paternal history which may have an impact on the outcome of this pregnancy.
- Fluarix, FluLaval, Fluarix Quadrivalent or FluLaval Quadrivalent vaccination including lot number and date of administration.
- Other drug/vaccine exposure including drug/vaccine name, route of administration, dose, lot number, indication and date of administration.
- Occurrence of AEs (if any), including onset/end date, outcome and relationship to GSK products.
- Name of HCP supervising pregnancy and contact information, if available.
- Any additional data that seems relevant for this study.

# 9.3.2.2. Questionnaire for pregnancy outcome data collection (Amended on 27 October 2017)

The following follow-up data will be collected using the questionnaire for <u>pregnancy</u> outcome data collection (i.e. Pregnancy Outcome Form):

- Pregnancy outcome.
- Method of delivery.
- Fetal/neonatal status, including description of birth defects if applicable.
- Infant information including gestational weeks at birth/miscarriage/termination, gender, length, weight, Apgar score.
- Additional drug/vaccine exposure including drug/vaccine name, route of administration, dose, lot number, indication and date of administration.
- AEs experienced by the fetus/infant or the mother.
- Name of the HCP supervising the infant and contact information, if available.
- Any additional data that seems relevant for this study.

#### 9.3.2.3. Questionnaire for infant data collection

The following data on the infant will be collected using the questionnaire for 6- and 12-month after delivery follow-up data collection (i.e. 6 and 12-month post-delivery Follow-Up Form):

- Infant status, including description of birth defects not diagnosed at the time of the initial follow-up, if applicable.
- AEs experienced by the infant.
- Additional drug/vaccine exposure including drug/vaccine name, route of administration, dose, lot number, indication and date of administration.
- Any additional data that seems relevant for this study.

## 9.4. Data sources (Amended on 27 October 2017)

Reporting of vaccine-exposed pregnancies to the Registry is voluntary. *Registration* can be initiated from a HCP, their staff or from a consumer. Permission from consumers is requested to obtain confirmation and follow-up from their HCP, as well as follow-up from the HCP participating in the care of the infant. A toll-free telephone number for reporting AEs and vaccine-exposed pregnancies to the Registry are listed in the product information leaflets and on the GSK Registry website. Retrospective post-marketing reports and relevant scientific publications are potential sources of additional information.

# 9.5. Study size

No minimum sample size is required for this *registry* study.

Refer to Section 9.2.1.2 for the size of the potential "at-risk" population and the number of pregnant vaccinees.

## 9.6. Data management

#### 9.6.1. Data collection (Amended on 27 October 2017)

Initial and follow-up data will be collected using 3 questionnaires. Initial data will be collected before the outcome is known. Follow-up of cases is performed at the following timepoints:

#### For consumer reports:

• At initial notification of pregnancy exposure: 2 attempts at 4-6 week intervals will be made to obtain more information about the pregnancy (e.g. estimated time of delivery (EDD) and/or last menstrual period (LMP) and to obtain permission to contact the patient's HCP

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

- Within 2 months after EDD: 1 additional attempt is made, if permission to contact the patient's HCP has not already been granted, to obtain more information about the pregnancy and obtain the permission to contact the patient's HCP.
- Within 2 months after EDD (and if the patient has not previously provided the contact information for her infant's HCP): 2 attempts at 4-6 week intervals will be made for all live births to obtain the contact information of the HCP supervising the health of the infant.

## For HCP reports:

• At initial notification of pregnancy exposure or once permission has been granted for reports initially received from a consumer, 2 attempts at 4-6 week intervals will be made to obtain more information via pregnancy follow-up form.

## For all reports:

- Within 2 months of the EDD, to ascertain outcome. *Two* attempts to obtain outcome information will be made before any case is considered lost to follow-up.
- An additional follow-up will be done for all live births (as confirmed around EDD) at approximately 6 months after the EDD to ascertain the presence of birth defects not diagnosed at the time of the initial follow-up. For this follow-up, the HCP supervising the health of the infant will be contacted.
- The last follow-up will be done *for all live births (as confirmed around EDD) at* approximately 12 months after the EDD to ascertain the presence of birth defects not diagnosed at previous follow-ups. *This follow-up will be done regardless of whether or not follow-up information was received at approximately 6 months after the EDD. For this follow-up, the HCP supervising the health of the infant will be contacted.*

# 9.6.2. Processing of reports (Amended on 27 October 2017)

Reports are entered into the GSK safety database by *the GSK Case Management Group responsible for all case entry into GSK's worldwide safety database* using existing mechanisms and practices. Follow-up is conducted by the Case Management Group.

The HCP supervising the pregnancy is contacted if she/he requests or if initial information is insufficient or needs clarification. The HCP supervising the health of the infant (and/or their staff) is contacted for all live births and if permission has been granted by the mother.

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

#### 9.6.2.1. Solicitation of outcomes (Amended on 27 October 2017)

As explained in section 9.6.1, within two months after the EDD and if the HCP has not already provided the outcome, she/he is sent a pregnancy outcome form (questionnaire). The mode of communication is generally via a standard letter.

Two attempts are made to secure the outcome information from the HCP. The second attempt also utilizes standard letter as mode of contact. For all live births (as confirmed around EDD) if the pregnant subject has previously provided her consent but has not already shared the contact information for the HCP supervising the health of the infant, two attempts are made to obtain this information.

For all live births (as confirmed around EDD) and with the mother's permission, two attempts are made to solicit information from the pediatrician and/or other specialists who have provided healthcare/consultation to the child up until 12 months of age (one attempt at around 6 months after EDD and another attempt at around 12 months after EDD).

#### 9.6.2.2. Classification of outcomes

This Registry uses the term 'birth defects' for outcomes sometimes referred to as 'congenital anomalies'. For purposes of analysis, pregnancy outcomes are dichotomized according to the presence or absence of birth defects. The latter group is further categorized as: 1) live births, 2) spontaneous abortions (i.e., pregnancy losses) and 3) induced abortions.

This Registry adopts a definition of a child with a birth defect as any live or stillborn neonate with a structural or chromosomal abnormality diagnosed before 6 years of age. The Registry employs a conservative approach of including all morphologic anomalies, including minor ones, as birth defects. To provide consistency in the definitions of major defects in this Registry, CDC MACDP criteria are used for the classification of defects [CDC, 2008; Correa-Villasenor, 2003]. Some of the conditions excluded from the MACDP criteria for major structural defects may actually have major clinical, functional, or genetic significance. Therefore, minor malformations not appearing in the CDC Inclusion List may be classified as birth defects in this Registry. In addition, CDC guidelines disqualify as defects those findings that are present in infants delivered at less than 36 weeks of gestation and are attributable to prematurity itself, such as a patent ductus arteriosus or inguinal hernias. Infants with infectious conditions (e.g., neonatal sepsis) or isolated biochemical abnormalities (e.g., hyperbilirubinemia) are classified as being without birth defects unless there is a possibility that the condition reflects an unrecognized congenital abnormality. All other congenital abnormalities are included in the 'birth defects' category, regardless of whether the neonate is delivered alive, including structural defects in neonates delivered prior to 20 weeks of gestation or weighing less than 500 g.

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

## 9.7. Data analysis (Amended on 27 October 2017)

Pregnancy outcomes include spontaneous abortion (pregnancy loss before 22 weeks gestation), fetal deaths/stillbirths (loss at or after 22 weeks gestation), elective/therapeutic abortions and live births. Gestational weeks are counted from the date of the LMP. The second trimester is considered to begin at week 14 and the third trimester begins at week 28. The presence or absence of birth defects or other abnormalities is evaluated within each of the preceding outcome categories.

Pregnancy outcomes are stratified by the trimester of exposure, with an additional stratum for preconception exposure with no subsequent administration of vaccine during pregnancy. Receiving multiple administrations of GSK sIIV during a single pregnancy is unlikely; however, if this does occur, reports of multiple exposures during a pregnancy are classified by the earliest trimester of exposure.

The calculations of risk for birth defects are made by dividing the number of infants with birth defects by the total number of infants with and without birth defects. Since the presence of birth defects will be assessed around EDD and at approximately 6 and 12 months after the EDD (for all live births), the calculation of risk will be performed for two separate cohorts: 1). the risk of birth defects for all subjects who completed the outcome form at around EDD (regardless of whether they were lost-to-follow up afterwards) and 2). the risk of birth defects for all subjects reporting live births and who completed either or both the 6- and 12-month post-delivery follow-up forms.

The outcomes of the study will be assessed against known rates from an external reference group for the likelihood of a safety signal warranting further investigation. In each periodic and the final reports, the data will be analyzed for all GSK sIIVs pooled and for each of the 4 vaccines separately. The analyses will also include data collected cumulatively in each individual registry up to the initiation of the combined Registry for GSK sIIVs. *Individual reports of birth defects following vaccination with any of the GSK sIIVs will also be evaluated for causal assessments, as appropriate.* 

The majority of spontaneous abortions occur early in pregnancy [Wilcox, 1981; Wilcox, 1983; Ellish, 1996]. If spontaneous abortions were to be evaluated as an outcome of interest, it would be essential to enroll pregnancies as soon as possible after vaccination with GSK sIIV. Because enrollment and recognition of pregnancy would occur at various times, it would be virtually impossible to meaningfully evaluate the effects of GSK sIIV on pregnancy loss [Kennedy, 2004]. Therefore, spontaneous abortions without birth defects are excluded from the risk calculations.

The risk in the general population of all birth defects meeting CDC criteria is approximately 3% (1 of 33) of live births [CDC, 2013]. The estimated risk cited in the medical literature varies because of differences in case definitions, populations sampled and ascertainment methods. The Collaborative Prenatal Project, using a broader case definition and prospective ascertainment, reports a frequency of 5% to 7% [Chung, 1975]. Most major structural defects originate during the first trimester of pregnancy, which is the critical time for organogenesis [Niebyl, 2012]. For such defects, exposures occurring in the second or third trimester are not likely to be causally associated.

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

However, for the sake of completeness and to enable the assessment of possible increases in the frequency of birth defects, all defects will be included in the periodic summary reports of this Registry and stratified by trimester of exposure.

Criteria for review of a specific individual report include:

- Is the timing of the vaccination with GSK sIIVs commensurate with the ontogenetic development of the organ(s) affected by the abnormalities?
- Is there another known or likely cause (e.g., pre-existing genetic or chromosomal defect or exposure to a known teratogen)?
- Is the congenital abnormality not previously described (i.e., is it new to medical science)?
- Is there a unique constellation of defects (i.e., is there a new syndrome)?

Criteria for review of aggregate data include:

- Is there a deviation from the expected frequency of all defects indicating an increase in the overall risk of defects?
- Is there a deviation from the expected frequencies of individual defects?
- Is there uniqueness (e.g., a pattern) of the abnormalities that is suggestive of a common etiology?

Studies have shown the risk of spontaneous abortion is high early in pregnancy and decreases substantially from week 8 to week 28, yielding a cumulative estimated risk of 10% to 22% [Wilcox, 1981; Wilcox, 1983; Wilcox, 1988; Fenster, 1997; Windham, 1997; Khattak, 1999; Anderson, 2000; Osborn, 2000].

While the Registry is to be limited to prospective reports, some pregnancy exposures are reported after pregnancy outcome has been identified (retrospective reports). The Registry will capture retrospective reports, but these reports will not be included in the analyses of prospective reports. In general, retrospective notification of outcomes following exposure to drugs or vaccines is biased toward reporting the severe and unusual cases and is not reflective of the general experience with the drug. Information about the total number of exposed pregnancies, i.e., the pool of exposures from which the retrospective reports arise, is unknown; therefore, incidences of outcomes cannot be calculated from these data. A series of reported birth defects, however, can be analyzed to detect patterns of specific congenital abnormalities and can identify early signals of new vaccine-associated risks. A section of each periodic summary report, separate from the analysis of prospective reports, will describe all abnormal outcomes of retrospectively reported cases.

# 9.8. Quality control

Data will be recorded using questionnaires. Subject data necessary for analysis, follow-up and reporting will be entered/transmitted into a validated database or data system. Data management will be performed in accordance with applicable GSK standards.

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

To ensure compliance with Good Clinical Practice (GCP) and all other applicable guidelines and regulatory requirements, GSK may conduct a quality assurance audit. Regulatory agencies may also conduct a regulatory inspection of this study. Such audits/inspections can occur at any time during or after completion of the study.

#### 9.9. Limitations of the research methods

This Registry is a prospective *voluntary* study. Active enrollment of a valid internal comparison group is not possible. Therefore, background risks from existing, external systems (e.g., the National Birth Defects Prevention Network and the National Center for Health Statistics) are used. The potential limitations of comparisons between Registry and background data depends upon the event(s) being compared and will be discussed on an *ad hoc* basis in the relevant periodic Registry reports. In addition, variations in the year-to-year (or strain), resulting in differences in the safety profiles of the vaccines, remain a possible limitation.

Refer to Section 9.1.2 for other potential limitations of the study.

#### 10. PROTECTION OF HUMAN SUBJECTS

# 10.1. Regulatory and ethical considerations, including the informed consent process

The study will be conducted in accordance with the International Conference on Harmonization (ICH) Guideline for GCP or other applicable guidelines, all applicable subject privacy requirements and the guiding principles of the Declaration of Helsinki.

The study has been designed and will be conducted in accordance with the ICH Harmonized Tripartite Guideline for clinical investigation of medicinal products in the pediatric population (ICH E11) and all other applicable ethical guidelines.

GSK will obtain favorable opinion/approval to conduct the study prior to study start or will document that neither a favorable opinion nor an approval to conduct the study is needed.

Conduct of the study includes, but is not limited to, the following:

- Institutional Review Board review and favorable opinion/approval of study protocol and any subsequent amendments;
- Institutional Review Board review and favorable opinion/approval of waiver for documentation of informed consent.

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

# 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

Reporting of vaccine-exposed pregnancies to the Registry is voluntary. All reports received by the Registry will be entered into the GSK safety database and reported to regulatory authorities according to applicable regulations.

# 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS (AMENDED ON 27 OCTOBER 2017)

Study information from this protocol will be posted on publicly available clinical trial registers following finalization of the protocol and, whenever possible, before initiation of the study.

GSK plans to continue the Registry for a minimum of 5 years. Summary reports will be written annually and will be submitted with the Periodic Benefit-Risk Evaluation Report for each GSK sIIV. Each report will summarize the adverse pregnancy outcomes that have been identified since the previous report and will also summarize cumulative results since the inception of the individual Registry. A final report will be written and submitted to CBER after the 5<sup>th</sup> annual report. In each periodic and the final reports, the data will be analyzed for all GSK sIIVs pooled and for each of the 4 vaccines separately. The analyses will also include data collected cumulatively in each individual registry up to the initiation of the combined Registry for GSK sIIVs. After submission of the final report, GSK will continue the Registry pending CBER review of the report and determination whether the Registry can be discontinued.

Summary results of observational studies that are designed to inform the safety or effectiveness, including cost-effectiveness, of GSK vaccines/products as used in ordinary clinical practice are publicly registered within 8 months of completion of the analysis. GSK also aims to publish the results of these studies in the searchable, peer reviewed scientific literature; manuscripts are submitted within 18 months of the completion of the analysis.

#### 13. REFERENCES

American College of Obstetricians and Gynecologists (ACOG) Influenza vaccination during pregnancy. ACOG Committee Opinion No. 305. *Obstet Gynecol* 2004; 104: 1125-1126.

Anderson AN, Wohlfahrt J, Christens P, Olsen J, Melbye M. Maternal age and fetal loss: population based register linkage study. *BMJ* 2000; 320:1708-1712.

Centers for Disease Control and Prevention (CDC). General Recommendations on Immunization. Recommendations of the Advisory Committee on Immunization Practices and the American Academy of Family Physicians. *MMWR* 2002; 51 (RR2): 1-36.

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

Centers for Disease Control and Prevention (CDC). Women with smallpox vaccine exposure during pregnancy reported to the National Smallpox Vaccine Pregnancy Registry -- United States, 2003. *MMWR* 2003; 52: 386-388.

Centers for Disease Control and Prevention (CDC). Birth Defects and Genetic Diseases Branch 6-digit code for reportable congenital anomalies. Revised 2008. Available at http://www.cdc.gov/ncbddd/birthdefects/documents/MACDPcode0807.pdf Accessed 22 August 2013.

Centers for Disease Control and Prevention (CDC). Influenza Vaccination Coverage Among Pregnant Women-United States, 2010–11 Influenza Season. *MMWR* 2011; 60: 1078-1082.

Centers for Disease Control and Prevention (CDC). Recent Trends in Births and Fertility Rates Through December 2012. Available at

http://www.cdc.gov/nchs/data/hestat/births\_fertility\_december\_2012/births\_fertility\_december 2012.htm

Accessed 29 August 2013.

Centers for Disease Control and Prevention (CDC). Birth defects. Available at http://www.cdc.gov/ncbddd/birthdefects/index.html Accessed 22 August 2013.

Chung CS, Myrianthopoulos NC. Factors affecting risks of congenital malformations: Reports from the Collaborative Perinatal Project. *Birth Defects Original Article Series* 1975; 11(10): 1-22.

Correa-Villasenor A, Cragan J, Kucik J, O'Leary L, Siffel C, Williams L. The Metropolitan Atlanta Congenital Defects Program: 35 years of birth defects surveillance at the Centers for Disease Control and Prevention. *Birth Defects Research (Part A)* 2003; 67: 617-624.

Ellish NJ, Saboda K, O'Connor J, et al. A prospective study of early pregnancy loss. *Hum Reprod* 1996; 11: 406-412.

Fenster L, Hubbard AE, Windham GC, Waller KO, Swan SH. A prospective study of work-related physical exertion and abortion. *Epidemiology* 1997; 8: 66-74.

Fluarix PI, 2013. Available at http://us.gsk.com/products/assets/us\_fluarix.pdf Accessed 13 February 2014.

Fluarix Quadrivalent PI, 2013. . Available at http://www.fda.gov/downloads/BiologicsBloodVaccines/Vaccines/ApprovedProducts/UCM220624.pdf

FluLaval PI, 2013. Available at http://us.gsk.com/products/assets/us\_flulaval.pdf Accessed 13 February 2014.

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

FluLaval Quadrivalent PI, 2013. Available at

http://www.fda.gov/downloads/BiologicsBloodVaccines/Vaccines/ApprovedProducts/UCM366070.pdf

Accessed 13 February 2014.

Honein MA, Paulozzi LJ, Cragan JD, Correa A. Evaluation of selected characteristics of pregnancy drug registries. *Teratology* 1999; 60(6): 356-364.

Kennedy DL, Uhl K, Kweder SJ. Pregnancy exposure registries. *Drug Safety* 2004; 27: 215-228.

Khattak S, K-Moghtader G, McMartin K, Barrera M, Kennedy D, Koren G. Pregnancy outcome following gestational exposure to organic solvents. *JAMA* 1999; 281(12): 1106-1109.

Neuzil KM, GW Reed, EF Mitchel, L Simonsen, MR Griffin. Impact of influenza on acute cardiopulmonary hospitalizations in pregnant women. *Am J Epidemiol* 1998; 148: 1094-1102.

Niebyl JR and JL Simpson. Chapter 8: Drugs and environmental agents in pregnancy and lactation: embryology, teratology and epidemiology. In Gabbe: Obstetrics: Normal and problem pregnancies, 6<sup>th</sup> ed; 2012: Saunders (Elsevier) p. 141.

Osborn JF, Cattaruzza MS, Spinelli A. Risk of spontaneous abortion in Italy, 1978-1995, and the effect of maternal age, gravity, marital status and education. *Am J Epidemiol* 2000; 151: 98-105.

Shields KE, Galil K, Seward J, et al. Varicella vaccine exposure during pregnancy: Data from the first 5 years of the Pregnancy Registry. *Obstet Gynecol* 2001; 98: 14-19.

Wilcox AJ, Treloar AE, Sandler DP. Spontaneous abortion over time: comparing occurrence in two cohorts of women a generation apart. *Am J Epidemiol* 1981; 114(4): 548-553.

Wilcox AJ. Surveillance of pregnancy loss in human populations. *Amer J Industr Med* 1983; 4: 285-291.

Wilcox AJ, Weinberg CR, O'Connor JF, et al. Incidence of early loss of pregnancy. *New Engl J Med* 1988; 319: 189-194.

Windham GC, Von Behren J, Fenster L, Schaefer C, Swan SH. Moderate maternal alcohol consumption and risk of spontaneous abortion. *Epidemiology* 1997; 8: 509-514.

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

# **ANNEX 1** List of stand-alone documents

| No. | Document Reference No | Date | Title |
|---|---|---|---|
| 1 | 201476 (EPI-FLU-039 VS US PR) | 13-MAY-2014 | List of stand-alone documents |
| 2 | 201476 (EPI-FLU-039 VS US PR) | 13-MAY-2014 | ENCePP Checklist for study protocols |
| 3 | 201476 (EPI-FLU-039 VS US PR) | 13-MAY-2014 | Glossary of terms |
| 4 | 201476 (EPI-FLU-039 VS US PR) | 11-OCT-2017 | Amendments and administrative changes to the protocol |
| 5 | 201476 (EPI-FLU-039 VS US PR) | 13-MAY-2014 | Trademarks |
| 6 | 201476 (EPI-FLU-039 VS US PR) | 13-MAY-2014 | Protocol Sponsor Signatory Approval |

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

# **ANNEX 2 ENCePP Checklist for study protocols**

# **ANNEX 3** Glossary of terms

Adverse event:

Any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product, or temporally associated with a study procedure.

An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e., lack of efficacy), abuse or

misuse.

eTrack:

GSK Biologicals' tracking tool for clinical/epidemiological trials.

GSK seasonal Inactivated Influenza Vaccines (GSK sIIVs): Fluarix®/ FluLaval®/ Fluarix® Quadrivalent/ FluLaval® Ouadrivalent vaccines

Non-interventional (observational) Human Subject Research:

Studies where medicinal products, should they be administered, are prescribed in normal (routine) medical practice. No medical care or medical/scientific procedures as required in a research protocol are administered to participants except as part of routine medical care.

**Post-Authorization Safety Study (PASS):** 

A pharmaco-epidemiological study or a clinical trial carried out in accordance with the terms of the marketing authorization, conducted with the aim of identifying or quantifying a safety hazard relating to an authorized medicinal product. This includes all GSK sponsored non-interventional studies and clinical trials conducted anywhere in the world that are in accordance with the terms of the European marketing authorization and where the investigation of safety is the specific stated objective.

Note: The phrase 'In accordance with the terms of the European marketing authorization' means that the product is used according to the European label (e.g., within the recommended dose range, the approved formulation, indication etc.).

**Prospective study:** 

A study that looks ahead for outcomes, e.g., the development of a disease, during the study period and relates this to other factors such as a potential risk due to exposure or protection factor(s). The study usually involves taking a cohort of subjects and watching them
201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

over a period for one or more common outcomes of

interest.

**Protocol amendment:** The International Conference on Harmonization (ICH)

defines a protocol amendment as: 'A written description of a change(s) to or formal clarification of a protocol.' GSK Biologicals further details this to include a change to an approved protocol that affects the safety of subjects, scope of the investigation, study design, or scientific

integrity of the study.

**Research protocol:** A document that describes the objective(s), design,

methodology, statistical considerations and organization

of a study. The protocol usually also gives the

background and rationale for the study, but these could be

provided in other protocol referenced documents.

**Retrospective study:** A study that looks backward in time (e.g., at events that

occurred in the past; outcomes and exposure can no longer be influenced), usually using medical records, databases or interviews in order to address one or more

study objectives.

**Self-contained study:** Study with objectives not linked to the data of another

study.

**Study population:** Sample of population of interest.

**Subject:** Term used throughout the protocol to denote an

individual who has been contacted in order to participate or participates in the epidemiological study or a person about whom some medical information has been recorded

in a database.

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

# ANNEX 4 Amendments and administrative changes to the protocol

| GlaxoSmithKline Biologicals SA | | |
|---|---|---|
| Vaccines R & D Protocol Amendment 1 | | |
| eTrack study number and Abbreviated Title: | 201476 (EPI-FLU-039 | VS US PR) |
| Amendment number: | Amendment 1 Final | |
| Amendment date: | 27 October 2017 | |
| Co-ordinating author: | PPD | , Scientific Writer |
| Rationale/background for changes: | | |

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

The current protocol is being amended to correct the following:

#### **Data collection:**

- Corrections were made throughout the protocol to reflect current practices for data collection, that two and not three follow up attempts are made around EDD to ascertain the presence of birth defects.
- Follow-up questionnaires for all live births were not being sent at approximately 6 and 12 months after EDD to ascertain the presence of birth defects not diagnosed at around EDD, contrary to what was described in the protocol. The importance of this information is acknowledged and both 6- and 12-month follow-up attempts will be implemented prospectively via a new data collection form.
- Originally, pregnant subjects enrolled into the registry had to sign a consent form only when subjects registered themselves into the registry, and to allow GSK to contact their HCPs at around EDD. Now, HCPs who register their pregnant patients will be encouraged to provide these with the consent form. With this consent, the HCP supervising the health of the infant up can also be contacted until 12 months after delivery. The consent form for the registry has also been refined to attempt to obtain contact information on the infant's healthcare provider. This new consent form will be implemented for all prospective reports.

#### **Exclusion criterion:**

• According to the exclusion criterion detailed in section 9.2.6 for the original protocol, subjects should be excluded from the registry if prenatal tests exist at the time of enrollment suggesting either normal or abnormal results. Considering that most pregnancies in the US go through fetal ultrasounds by the first trimester of gestation, this exclusion criterion will pointedly limit the number of subjects who enroll into the registry and enrich for subjects with low prenatal care coverage. The registry protocol has been updated to reflect its current practices: pregnancies will be excluded from enrollment only if abnormal pregnancy outcomes are diagnosed before receipt of a GSK seasonal influenza vaccine.

#### **Pregnancy registry reports:**

• The dates for submission of the annual reports have been updated to reflect newer PBRER submission dates.

# Post-marketing exposure in pregnant women:

• Numbers and outcomes of women exposed to each GSK sIIV during pregnancy since their respective launches and spontaneously reported into our safety database worldwide were updated.

# **Data Analysis:**

• Since the 6- and 12-month follow-ups will only be done prospectively, we propose calculating the risk of birth defects for two separate cohorts: 1). the risk of birth defects for all mother-child pairs with complete pregnancy outcome forms at around EDD (regardless of whether they were lost-to-follow up afterwards) and 2). the risk of birth defects for all mother-child pairs reporting live births at around EDD and who completed either or both the 6- and 12-month post-delivery follow-up forms.

Since this registry is currently ongoing, changes beyond those related to the items above were limited to minor updates for clarity purposes.

These changes will be implemented within 30 days of approval by the FDA.

Amended text has been included in *bold italics* and deleted text in <del>strikethrough</del> in the following sections:

# Cover page:

| Authors | , Safety Scientist, |
|---|---|
| | Safety Evaluation & Risk Management,<br>Vaccine Clinical Safety and<br>Pharmacovigilance |
| | • PPD , Head, Safety Evaluation & Risk Management, Vaccine Clinical Safety and Pharmacovigilance |
| | • PPD , Local Medical Lead |
| | • PPD , Clinical and Epidemiology Project Lead, Influenza Vaccines |
| | • PPD , Regulatory Affairs |
| | • PPD , Manager, CMG |
| | • PPD , Clinical Safety Associate |
| | • PPD , Director, CMG |
| | • PPD , Study Delivery Lead |
| | • PPD , Senior Epidemiology<br>Expert, US RDC |
| | • PPD , Lead Epidemiologist |

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

Copyright 2014 of the GlaxoSmithKline group of companies. All rights reserved. Unauthorized copying or use of this information is prohibited

© [2014-2017] GSK group of companies or its licensor

#### **Synopsis:**

# Study design

- This study is a transition of existing ongoing pregnancy registries for *Fluarix*, *FluLaval* and *Fluarix Quadrivalent* and an ongoing PASS for *FluLaval Quadrivalent* into a combined PASS for these four GSK sIIVs.
- This is an exploratory prospective, observational, cohort study. The GSK sIIVs pregnancy registry study requires voluntary, prospective\* reporting of eligible pregnancies by patients and healthcare professionals (HCPs). Data such as vaccination with GSK sIIVs during pregnancy or within 28 days preceding conception, potential confounding factors (such as exposure to other medications) and information related to the outcome of the pregnancy will be collected prospectively.

\*Some pregnancy exposures may be reported when the outcome is unknown (prospective reports).

Some pregnancy exposures may be reported after pregnancy outcome has been identified (retrospective reports). The Registry will capture retrospective reports, but these reports will not be included in the analyses of prospective reports.

- This study is a post-marketing commitment in the US.
- Study population: pregnant women, vaccinated with GSK sIIVs during pregnancy or within 28 days preceding conception volunteering to take part in the study.
- Type of study: self-contained.
- Data collection: initial and follow-up data will be collected using questionnaires (Registration Initial notification form, Pregnancy Outcome form and 6 and 12-month post-delivery follow-up form). Initial data can be collected from pregnant subjects, their healthcare providers or both. Follow-up of cases is performed within 2 months of the estimated date of delivery (EDD) to ascertain outcome and approximately 6 months and 12 months after the EDD (for all live births for whom the contact details of their HCP will be available) to ascertain the presence of birth defects not diagnosed before. Follow-up questionnaires can only be completed by healthcare providers and/or HCP staff

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

participating in the care of the pregnant female or offspring, as applicable.

• After transition of the ongoing pregnancy registries into one combined PASS for GSK sIIVs, data will be collected for a minimum of 5 years starting Q2 2014

Population, including the setting and study population

In the US, GSK sIIVs are indicated for prevention of disease caused by influenza A subtype viruses and type B viruses contained in the vaccine. GSK sIIVs are approved for use in persons 3 years of age and older. Currently, GSK sIIVs are approved for use in persons 3 years of age and older or 6 months of age and older, depending on the vaccine.

# Size of the potential "at-risk" population

In the year 2012, the fertility rate in the US was 63.2 births per 1000 women aged 15-44 years and there were 3.96 million births [CDC, 2012].

# Number of pregnant vaccinees

Although the number of pregnant women who will be vaccinated with GSK IIVs *through this registry* is impossible to predict, experiences with other vaccine pregnancy registries indicate that it is likely that fewer than 100 pregnancies per year will be registered for each of the vaccines.

**Data sources** 

Reporting of vaccine-exposed pregnancies to the Registry is voluntary. Registration can be initiated from a HCP or from a consumer in the latter case. Permission *from consumers* is requested to obtain confirmation and follow-up from their HCP, *as well as follow-up from the HCP of their infant*. A toll-free telephone number for reporting adverse events (AEs) and vaccine-exposed pregnancies to the Registry are listed in the product information leaflet and on the GSK Registry website. Retrospective post-marketing reports and relevant scientific publications are potential sources of additional information.

# Data analysis

Pregnancy outcomes include spontaneous abortion (pregnancy loss before 20 22 weeks gestation), fetal deaths/stillbirths (loss at or after 20 22 weeks gestation), elective/therapeutic abortions and live births. The presence or absence of birth defects or other abnormalities is evaluated within each of the preceding outcome categories.

Pregnancy outcomes are stratified by the trimester of exposure, with an additional stratum for preconception exposure with no subsequent administration of vaccine

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

during pregnancy. Reports of multiple exposures during a pregnancy are classified by the earliest trimester of exposure. The calculations of risk for birth defects are made by dividing the number of infants with birth defects by the total number of infants with and without birth defects. An exact 95% confidence interval is calculated using standard statistical software. The outcomes of the study will be assessed against known rates from an external reference group for the likelihood of a safety signal warranting further investigation.

Spontaneous abortions without birth defects are excluded from the risk calculations.

All defects regardless of trimester of vaccine exposure will be included in the periodic summary reports of this Registry and stratified by trimester of exposure.

A section of each periodic summary report, separate from the analysis of prospective reports, will describe all abnormal outcomes of retrospectively reported cases.

Milestones

Summary reports with cumulative analyses will be written annually and submitted with the Periodic Benefit-Risk Evaluation Report (PBRER) for each GSK sIIV. A final report will be written and submitted 18 months after the last annual report. A final report will be written and submitted 18 months after the last annual report.

After submission of the final report, GSK will continue the Registry pending Center for Biologics Evaluation and Research (CBER) review of the report and determination whether the Registry can be discontinued.

# **Section 6** Milestones

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

| Milestone | Planned date <sup>a</sup> |
|---|---|
| Start of data collection | 01 June 2014 <sup>b</sup> |
| End of data collection | 31 May 2019 ° |
| Annual report 1 (2014-2015 influenza season) | 10 February 2016 30 June 2015 |
| Annual report 2 (2015-2016 influenza season) | 10 February 2017 30 June 2016 |
| Annual report 3 (2016-2017 influenza season) | 10 February 2018 30 June 2017 |
| Annual report 4 (2017-2018 influenza season) | 10 February 2019 30 June 2018 |
| Annual report 5 (2018-2019 influenza season) | <del>30 June 2019-10 February 2020</del> |
| Final report | August 2021 06 March 2020 |

<sup>&</sup>lt;sup>a</sup> The *Fluarix* and *FluLaval* Registries were originally initiated on 02 Sep 2011. The *Fluarix Quadrivalent* and *FluLaval Quadrivalent* Registries were originally initiated on 30 Aug 2013 and 30 Nov 2013, respectively. *In* **2014**. the ongoing Registries will be were combined and converted into a PASS. GSK plans to continue the Registry for a minimum of 5 years, starting Q2 2014.

# **Section 7.1.1.2 Post marketing exposure in pregnant women**

<sup>&</sup>lt;sup>b</sup> Women vaccinated with GSK sIIVs during pregnancy or within 28 days preceding conception, reported before the planned date of start of data collection (01 June 2014) but for which the pregnancy outcome is not yet known, may be enrolled retroactively in the Registry.

<sup>&</sup>lt;sup>c</sup> After submission of the final report, GSK will continue the Registry pending Center for Biologics Evaluation and Research (CBER) review of the report and determination whether the Registry can be discontinued.

#### Fluarix:

Overall, as of 31 August 2013 31 May 2017, GSK had received 243 236 reports of exposure to *Fluarix* during pregnancy since its launch on 04 July 1991. The outcomes of the 243 236 pregnancies are summarized in Table 2.

Table2 Outcomes of pregnancy exposed to Fluarix

| Outcome | Number of Cases since launch (n) |
|---|---|
| Live infant, no apparent congenital anomaly * | <del>55</del> <b>52</b> |
| Live infant with congenital anomaly | 4 1 |
| Elective termination, no apparent congenital anomaly * | 4 0 |
| Elective termination with congenital anomaly | 21 |
| Spontaneous abortion, no apparent congenital anomaly * | <del>12</del> 8 |
| Spontaneous abortion with congenital anomaly | 0-1 |
| Stillbirth, no apparent congenital anomaly * | 20 |
| Stillbirth with congenital anomaly | 4 0 |
| Ectopic pregnancy | 0 |
| Molar pregnancy | 0 |
| Pregnancy ongoing, lost to follow-up or unknown | <del>166-</del> 173 |
| Total | <del>243</del> <b>236</b> |

<sup>\*</sup> Pregnancy outcome categories stating no apparent congenital anomaly include outcomes where it is unknown whether a congenital anomaly occurred.

# FluLaval:

Overall, as of 17 December 2013 31 May 2017, GSK had received 128 130 reports of exposure to FluLaval during pregnancy since launch on 18 December 1992. The outcomes of the 128 130 pregnancies are summarized in Table 3.

Table 3 Outcomes of pregnancy exposed to FluLaval

| Outcome | Number of Cases since launch |
|---|---|
| Live Infant, no apparent congenital anomaly * | <del>26</del> <b>46</b> |
| Live infant with congenital anomaly | 21 |
| Elective termination, no apparent congenital anomaly* | 0 |
| Elective termination with congenital anomaly | 0 |
| Spontaneous abortion, no apparent congenital anomaly* | 3 |
| Spontaneous abortion with congenital anomaly | 0 |
| Stillbirth, no apparent congenital anomaly* | 0 |
| Stillbirth with congenital anomaly | 0 |
| Ectopic pregnancy | 0 |
| Molar pregnancy | 0 |
| Pregnancy ongoing / Unknown / Lost to Follow-up | <del>97</del> <b>80</b> |
| Not applicable | 0 |
| Total | <del>128</del> <b>130</b> |

<sup>\*</sup> Pregnancy outcome categories stating no apparent congenital anomaly include outcomes where it is unknown whether a congenital anomaly occurred.

# Section 7.1.2.2 Post marketing exposure in pregnant women

Fluarix Quadrivalent:

Overall, as of 19 February 2014 31 May 2017, GSK had received 25 64 reports of exposure to Fluarix Quadrivalent during pregnancy since launch on 5 August 2013. The outcomes of the 64 pregnancies are summarized in Table 4.

Table 4 Outcomes of pregnancy exposed to Fluarix Quadrivalent

| Outcome | Number of Cases since launch (n) |
|---|---|
| Live infant, no apparent congenital anomaly * | 15 |
| Live infant with congenital anomaly | 0 |
| Elective termination, no apparent congenital anomaly * | 0 |
| Elective termination with congenital anomaly | 0 |
| Spontaneous abortion, no apparent congenital anomaly * | 1 |
| Spontaneous abortion with congenital anomaly | 1 |
| Stillbirth, no apparent congenital anomaly * | 0 |
| Stillbirth with congenital anomaly | 0 |
| Ectopic pregnancy | 0 |
| Molar pregnancy | 0 |
| Pregnancy ongoing, lost to follow-up or unknown | 47 |
| Total | 64 |

Of the 25 pregnancy reports, 22 were ongoing at the time of reporting and 3 were considered lost to follow up.

FluLaval Quadrivalent:

Overall, as of 17 December 2013 31 May 2017, GSK had received 5 8 reports of exposure to FluLaval Quadrivalent during pregnancy since launch on 15 August 2013. At the time of the reporting, all 5 8 pregnancies were ongoing or lost to follow-up.

#### Section 7.1.3 Medical conditions for use

The GSK sIIVs are approved by the US Food and Drug Administration (FDA) for prevention of disease caused by influenza A subtype viruses and type B viruses contained in the vaccines (Table 5). In the US, the GSK sIIVs are approved for use in persons 3 years of age and older or 6 months of age and older, depending on the vaccine.

# **Section 7.2** Rationale

The purpose of this pregnancy registry study is to detect and describe abnormal pregnancy outcomes in women intentionally or unintentionally vaccinated with any of the four GSK sIIVs. The combination of the large number of women who are of reproductive capacity in the indicated age range for vaccination with GSK sIIVs, and the lack of data concerning vaccination during pregnancy, makes such a Registry an important

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

component of the ongoing program to assess the safety of these vaccines. This study is a transition of existing ongoing pregnancy registries for *Fluarix*, *FluLaval*, and *Fluarix Quadrivalent* and an ongoing PASS for *FluLaval Quadrivalent* into a combined PASS for GSK sIIVs. Timelines for collection of follow up data will be adapted in order to correspond to the follow-up timelines of other GSK pregnancy registries.

The Registry requires voluntary, prospective reporting of eligible pregnancies by patients and healthcare professionals (HCPs). Patient confidentiality is strictly maintained. The intent of the Registry is to prospectively collect data such as vaccination with any of the four GSK sIIVs during pregnancy or within 28 days preceding conception, potential confounding factors (such as exposure to other medications) and information related to the outcome of the pregnancy.

The GSK sIIV pregnancy registry study will be maintained by GSK's Vaccine Clinical Safety and Pharmacovigilance (VCSP) department.

# Section 9.1.1 Study design overview

• Data collection: initial and follow-up data will be collected using 2 3 questionnaires. *Data for enrollment will be collected using the Initial Notification Form.* Follow-up of cases is performed within 3 2 months of the estimated date of delivery (EDD) to ascertain *pregnancy* outcome (through the *Pregnancy Outcome Form*) and approximately 6 months and 12 months after the EDD (for all live births for whom the contact details of their HCP will be available) to ascertain the presence of birth defects not diagnosed before (through the 6- and 12-month post-delivery Follow-Up Form).

#### Section 9.1.2 Rationale for the study design

This study is designed as a *condition based* Registry *as opposed to a disease registry*. After market authorization, adverse events (AEs) that occur after administration of the vaccine can and should always be reported. In that case, however, there is no clear group in which the events occur and so a proper rate of occurrence cannot be estimated. In this pregnancy registry, participants are recruited between administration of the vaccine and the potential occurrence of an AE (i.e., a teratogenic effect in the offspring). This allows for a more proper estimation of the rate of occurrence of these events. Nevertheless, the results of this study still need to be regarded with caution as the exact number of women exposed during pregnancy is unknown. Incidences of events cannot therefore be calculated from the study data.

Furthermore, it is likely that pregnant women who accept vaccination may differ from those who refuse vaccination in underlying health status, propensity to seek medical care, propensity to report AEs and differences in access to medical care in general. The differential response/participation by vaccinated versus unvaccinated pregnant women in a pregnancy registry could significantly bias risk estimates and possibly in unpredictable ways, because of the inability to collect adequate data to characterize the non-responders.

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

Therefore, the risks of any identified birth defects will be compared to those in the general population, such as that defined by the Metropolitan Atlanta Congenital Defects Program (MACDP).

# **Section 9.2.1.1** Patient population

In the US, the GSK sIIVs are indicated for prevention of disease caused by influenza A subtype viruses and type B viruses contained in the vaccine. GSK sIIVs are approved for use in persons 3 years of age and older or 6 months of age and older, depending on the vaccine.

The study population includes women vaccinated with any of the four GSK sIIVs during pregnancy or within 28 days preceding conception.

# **Section 9.2.1.2 Potential annual exposure**

# Number of pregnant vaccinees

The four GSK sIIVs are classified as Pregnancy Category B. Although the number of pregnant women who will be vaccinated with GSK sIIV *with this registry* is impossible to predict, experiences with other vaccine pregnancy registries (e.g., smallpox vaccine [CDC, 2003], varicella vaccine [Shields, 2001] and *Twinrix*) indicate that it is likely that fewer than 100 pregnancies per year will be registered for each of the vaccines.

#### Section 9.2.2 Patient recruitment

Reporting of vaccine-exposed pregnancies to the Registry is voluntary. Reporters become aware of the Registry through the US Prescribing Information (PI) and *in the case of healthcare providers* the GSK Registry website. The PIs for each of the sIIVs and GSK *registry* website each give a brief summary of the purpose and intent of the Registry, along with telephone and fax contact information. *The forms for enrolling and reporting outcomes are also accessible to healthcare providers through the GSK Registry website*. Additionally, GSK has requested that information regarding GSK pregnancy registries be posted directly on the FDA website.

# Section 9.2.5 Inclusion criteria

A subject will be included in the Registry if all of the following criteria are met:

- Exposure to GSK sIIVs occurs during pregnancy or within 28 days preceding conception.
- Subject is a US resident.
- A HCP is identified (name, address and phone number).
- Subject can be identified (by GSK or HCP).

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

Data from registered subjects will be included in the analyses if the following criterion is met:

• Pregnancy is ongoing and the outcome is unknown at the time of initial report.

#### Section 9.2.6 Exclusion criteria

Data from registered subjects will not be included in the analyses if the following criterion is met:

• Outcome of pregnancy is known at the time of initial report. Types of known outcomes include prenatal testing reports in which the results are abnormal or outside the reference range, indicating possible abnormality in the fetus. Pregnancies in which prenatal testing indicates a normal pregnancy would also be excluded because inclusion of such pregnancies could potentially bias results toward a lower overall estimate of risk for defects [Honein, 1999]. Typically pregnancies > 16 weeks gestation will have undergone prenatal testing that can identify whether a child has congenital abnormalities.

# Section 9.3.2 Data to be collected

Data will be collected using 2 3 questionnaires; one for enrollment (i.e. Initial Notification Form) initial data and, one for follow-up data after the EDD (i.e. Pregnancy Outcome Form) and one for infant data at about 6 and 12 months after EDD (i.e. 6- and 12-month post-delivery Follow-Up Form.

With the information gathered from these questionnaires, the frequency of birth defects among enrolled subjects will be calculated and individual reports will be evaluated for causal assessments, if possible.

#### Section 9.3.2.1 Questionnaire for initial data collection

The following initial data will be collected using the questionnaire for initial data collection (i.e. Initial Notification Form):

- Patient identifier.
- Maternal medical and family history including date of birth, date of last menstrual period (LMP), EDD, ethnicity.
- Type of conception.
- Prenatal testing.
- Number and outcome of previous pregnancies, including details of birth defects if applicable.
- Maternal/paternal history which may have an impact on the outcome of this pregnancy.

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

- Fluarix, FluLaval, Fluarix Quadrivalent or FluLaval Quadrivalent vaccination including lot number and date of administration.
- Other drug/vaccine exposure including drug/vaccine name, route of administration, dose, lot number, indication and date of administration.
- Occurrence of AEs (if any), including onset/end date, outcome and relationship to GSK products.
- Name of HCP name supervising pregnancy and contact information, if available.
- Any additional data that seems relevant for this study.]

# Section 9.3.2.2 Questionnaire for follow-up pregnancy outcome data collection

The following follow-up data will be collected using the questionnaire for follow-up pregnancy outcome data collection (i.e. Pregnancy Outcome Form):

- Pregnancy outcome.
- Method of delivery.
- Fetal/neonatal status, including description of birth defects if applicable.
- Infant information including gestational weeks at birth/miscarriage/termination, gender, length, weight, Apgar score.
- Additional drug/vaccine exposure including drug/vaccine name, route of administration, dose, lot number, indication and date of administration.
- AEs experienced by the fetus/infant or the mother.
- *Name of the HCP name supervising the infant* and contact information.
- Any additional data that seems relevant for this study.

# Section 9.3.2.3 Questionnaire for infant data collection

The following data on the infant will be collected using the questionnaire for 6- and 12-month after delivery follow-up data collection (i.e. 6 and 12-month post-delivery Follow-Up Form):

- Infant status, including description of birth defects not diagnosed at the time of the initial follow-up, if applicable.
- AEs experienced by the infant.
- Additional drug/vaccine exposure including drug/vaccine name, route of administration, dose, lot number, indication and date of administration.
- Any additional data that seems relevant for this study.

# Section 9.4 Data sources

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

Reporting of vaccine-exposed pregnancies to the Registry is voluntary. Registration can be initiated from a HCP or from a consumer; in the latter case permission is requested to obtain confirmation and follow-up from their HCP. Registration can be initiated from a HCP, their staff or from a consumer. Permission from consumers is requested to obtain confirmation and follow-up from their HCP, as well as follow-up from the HCP participating in the care of the infant. A toll-free telephone number for reporting AEs and vaccine-exposed pregnancies to the Registry are listed in the product information leaflets and on the GSK Registry website. Retrospective post-marketing reports and relevant scientific publications are potential sources of additional information.

# Section 9.5 Study size

No minimum sample size is required for this descriptive registry study.

Refer to Section 9.2.1.2 for the size of the potential "at-risk" population and the number of pregnant vaccinees.

#### Section 9.6.1 Data collection

Initial and follow-up data will be collected using 2 *3* questionnaires. Initial data will be collected before the outcome is known. Follow-up of cases is performed at the following timepoints:, with each follow-up independent from the others:

#### For consumer reports:

- At initial notification of pregnancy exposure: 2 attempts at 4-6 week intervals will be made to obtain more information about the pregnancy (e.g. estimated time of delivery (EDD) and/or last menstrual period (LMP) and to obtain permission to contact the patient's HCP
- Within 2 months after EDD, 1 additional attempt is made, if permission to contact the patient's HCP has not already been granted, to obtain more information about the pregnancy and obtain the permission to contact the patient's HCP.

# For HCP reports:

• At initial notification of pregnancy exposure or once permission has been granted for reports initially received from a consumer, 2 attempts at 4-6 week intervals will be made to obtain more information via pregnancy follow-up form. If the HCP submitting the report (or his/her staff) participating in the care of the pregnant female, reports will only be processed if contact information for the relevant HCP supervising the pregnancy is provided and/or if permission has been granted by the mother.

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

- Within 3 2 months of the EDD, to ascertain outcome. At least three *Two* attempts to obtain outcome information will be made before any case is considered lost to follow-up.
- An additional follow-up will be done for all live births (as confirmed around EDD) approximately 6 months after the EDD to ascertain the presence of birth defects not diagnosed at the time of the initial follow-up.
- The last follow-up will be done *for all live births (as confirmed around EDD) at* approximately 12 months after the EDD to ascertain the presence of birth defects not diagnosed at previous follow-ups.

# Section 9.6.2 Processing of reports

Initial rReports are entered into the GSK safety database by Client Response Center staff GSK Case management group responsible for all case entry into GSK's worldwide safety database using existing mechanisms and practices. Follow-up is conducted by the Case Management Group. The HCP supervising the pregnancy is contacted if she/he requests or if initial information is insufficient or needs clarification. The HCP supervising the health of the infant (and/or their staff) is contacted for all live births and if permission has been granted by the mother. The HCP is encouraged to keep a copy of the initial completed form in the patient's chart.

#### Section 9.6.2.1 **Solicitation of outcome**

As explained in section 9.6.1, within three two months after the EDD and if the HCP has not already provided the outcome, she/he is sent an a pregnancy outcome form (questionnaire), along with a copy of the initial completed pregnancy form. The mode of communication is the one through which the initial information was received (telephone, fax, or postal mail) generally via a standard letter.

At least three *Two* attempts are made to secure the outcome information from the HCP. The second and third attempt *also* utilizes *standard letter as mode* all modes of contact available (mail, fax, telephone). If outcome is not received from the HCP and contact information is available for the patient, she is then contacted by mail or fax. In the event of an abnormal outcome *For all live births (as confirmed around EDD)* and with the mother's permission, attempts are made to solicit information from the pediatrician and/or other specialists who have provided healthcare/consultation to the child up *until 12 months of age*.

# Section 9.7 Data analysis

Pregnancy outcomes include spontaneous abortion (pregnancy loss before 20 22 weeks gestation), fetal deaths/stillbirths (loss at or after 20 22 weeks gestation), elective/therapeutic abortions and live births. Gestational weeks are counted from the date of the LMP. The second trimester is considered to begin at week 14 and the third

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

trimester begins at week 28. The presence or absence of birth defects or other abnormalities is evaluated within each of the preceding outcome categories.

Pregnancy outcomes are stratified by the trimester of exposure, with an additional stratum for preconception exposure with no subsequent administration of vaccine during pregnancy. Receiving multiple administrations of GSK sIIV during a single pregnancy is unlikely; however, if this does occur, reports of multiple exposures during a pregnancy are classified by the earliest trimester of exposure.

The calculations of risk for birth defects are made by dividing the number of infants with birth defects by the total number of infants with and without birth defects. Since the presence of birth defects will be assessed around EDD and at approximately 6 and 12 months after the EDD (for all live births), the calculation of risk will be performed for two separate cohorts: 1). the risk of birth defects for all subjects who completed the outcome form at around EDD (regardless of whether they were lost-to-follow up afterwards) and 2). the risk of birth defects for all subjects reporting live births and who completed either or both the 6- and 12-month post-delivery follow-up forms.

The outcomes of the study will be assessed against known rates from an external reference group for the likelihood of a safety signal warranting further investigation. In each periodic and the final reports, the data will be analyzed for all GSK sIIVs pooled and for each of the 4 vaccines separately. The analyses will also include data collected cumulatively in each individual registry up to the initiation of the combined Registry for GSK sIIVs. *Individual reports of birth defects following vaccination with any of the GSK sIIVs will also be evaluated for causal assessments, as appropriate.* 

The majority of spontaneous abortions occur early in pregnancy [Wilcox, 1981; Wilcox, 1983; Ellish, 1996]. If spontaneous abortions were to be evaluated as an outcome of interest, it would be essential to enroll pregnancies as soon as possible after vaccination with GSK sIIV. Because enrollment and recognition of pregnancy would occur at various times, it would be virtually impossible to meaningfully evaluate the effects of GSK sIIV on pregnancy loss [Kennedy, 2004]. Therefore, spontaneous abortions without birth defects are excluded from the risk calculations.

The risk in the general population of all birth defects meeting CDC criteria is approximately 3% (1 of 33) of live births [CDC, 2013]. The estimated risk cited in the medical literature varies because of differences in case definitions, populations sampled and ascertainment methods. The Collaborative Prenatal Project, using a broader case definition and prospective ascertainment, reports a frequency of 5% to 7% [Chung, 1975]. Most major structural defects originate during the first trimester of pregnancy, which is the critical time for organogenesis [Niebyl, 2012]. For such defects, exposures occurring in the second or third trimester are not likely to be causally associated. However, for the sake of completeness and to enable the assessment of possible increases in the frequency of birth defects, all defects will be included in the periodic summary reports of this Registry and stratified by trimester of exposure.

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

Criteria for review of a specific individual report include:

- Is the timing of the vaccination with GSK sIIVs commensurate with the ontogenetic development of the organ(s) affected by the abnormalities?
- Is there another known or likely cause (e.g., pre-existing genetic or chromosomal defect or exposure to a known teratogen)?
- Is the congenital abnormality not previously described (i.e., is it new to medical science)?
- Is there a unique constellation of defects (i.e., is there a new syndrome)?

Criteria for review of aggregate data include:

- Is there a deviation from the expected frequency of all defects indicating an increase in the overall risk of defects?
- Is there a deviation from the expected frequencies of individual defects?
- Is there uniqueness (e.g., a pattern) of the abnormalities that is suggestive of a common etiology?

Studies have shown the risk of spontaneous abortion is high early in pregnancy and decreases substantially from week 8 to week 28, yielding a cumulative estimated risk of 10% to 22% [Wilcox, 1981; Wilcox, 1983; Wilcox, 1988; Fenster, 1997; Windham, 1997; Khattak, 1999; Anderson, 2000; Osborn, 2000].

While the Registry is to be limited to prospective reports, some pregnancy exposures are reported after pregnancy outcome has been identified (retrospective reports). The Registry will capture retrospective reports, but these reports will not be included in the analyses of prospective reports. In general, retrospective notification of outcomes following exposure to drugs or vaccines is biased toward reporting the severe and unusual cases and is not reflective of the general experience with the drug. Information about the total number of exposed pregnancies, i.e., the pool of exposures from which the retrospective reports arise, is unknown; therefore, incidences of outcomes cannot be calculated from these data. A series of reported birth defects, however, can be analyzed to detect patterns of specific congenital abnormalities and can identify early signals of new vaccine-associated risks. A section of each periodic summary report, separate from the analysis of prospective reports, will describe all abnormal outcomes of retrospectively reported cases.

#### Section 9.9 Limitations of the research methods

This Registry is a prospective cohort study convenience sample of pregnant women who are followed prospectively. Active enrollment of a valid internal comparison group is not possible. Therefore, background risks from existing, external systems (e.g., the National Birth Defects Prevention Network and the National Center for Health Statistics) are used. The potential limitations of comparisons between Registry and background data depends upon the event(s) being compared and will be discussed on an ad hoc basis in the relevant periodic Registry reports. In addition, variations in the

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

year-to-year (or strain), resulting in differences in the safety profiles of the vaccines, remain a possible limitation.

Refer to Section 9.1.2 for other potential limitations of the study.

# **ANNEX 5** Trademarks

The following trademarks are used in the present study outline. Note: In the remainder of the document, the names of the vaccines will be written without the superscript symbol  $^{\text{TM}}$  or  $^{\text{R}}$ .

| Trademarks of the GSK group of companies |
|------------------------------------------|
| Fluarix <sup>®</sup> |
| Fluarix® Quadrivalent |
| FluLaval® |
| FluLaval <sup>®</sup> Quadrivalent |
| Twinrix <sup>®</sup> |

| Generic description |
|-------------------------------------------------------------|
| trivalent inactivated influenza virus vaccine |
| quadrivalent inactivated influenza virus vaccine |
| trivalent inactivated influenza virus vaccine |
| quadrivalent inactivated influenza virus vaccine |
| hepatitis A inactivated & hepatitis B (recombinant) vaccine |

201476 (EPI-FLU-039 VS US PR) Protocol Amendment 1 Final

# **ANNEX 6** Protocol Amendment 1 sponsor signatory approval

| eTrack study number and Abbreviated Title | 201476 (EPI-FLU-039 VS US PR) |
|---|---|
| Date of protocol | Amendment 1 Final: 27 October 2017 |
| Detailed Title | Fluarix®/FluLaval®/Fluarix® Quadrivalent/FluLaval® Quadrivalent Pregnancy Registry: a prospective, exploratory, cohort study to detect and describe abnormal pregnancy outcomes in women intentionally or unintentionally vaccinated with Fluarix® or Fluarix® Quadrivalent or FluLaval® or FluLaval® Quadrivalent during pregnancy or within 28 days preceding conception. |
| Sponsor signatory | Anne Yeakey, Head, Safety Evaluation & Risk Management, Vaccine Clinical Safety and Pharmacovigilance |
| Signature | |
| Date | |